CLINICAL TRIAL: NCT01283776
Title: A Phase II Study to Investigate the Efficacy of Cyclophosphamide as Sole Graft-Versus-Host-Prophylaxis After Allogeneic Stem Cell Transplantation
Brief Title: Cyclophosphamide as Sole Graft-Versus-Host-Prophylaxis After Allogeneic Stem Cell Transplantation
Acronym: OCTET-CY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Christoph Scheid, PD Dr. Christoph Scheid, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Uni-Koeln-1430
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Myeloma; Non-Hodgkin-Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment arm (Experimental): Cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — 100 mg/kg total dose, infused on day +3 and +3 after allogeneic stem cell transplantation

SUMMARY:
A phase II clinical study to assess the efficacy of post-transplantation cyclophosphamide as single-agent GvHD prophylaxis after allogeneic hematopoietic stem cell transplantation in patients with multiple myeloma or lymphoma and to describe the influence of the modified immunosuppression concept on relapse rates, minimal residual disease, immune reconstitution and chimerism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma, Non-Hodgkin's lymphoma or Hodgkin's disease after allogeneic stem cell transplantation with reduced intensity conditioning

  * Written informed consent
  * No uncontrolled infections

Exclusion Criteria:

* Severe organ dysfunction defined as:
* Cardiac left ventricular ejection fraction (LVEF) of less than 35%
* diffusing lung capacity (DLCO) of less than 40%
* total lung capacity (TLC) of less than 40%
* forced expiratory volume (FEV1) of less than 40%
* total bilirubin >3mg/dl
* creatinine-clearance of less than 40 ml/min
* pregnancy or breast feeding
* participation in other experimental drug trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of patients not requiring additional immunosuppression | day 100 after transplant
  The primary endpoint is met if at least 1 of the 5 first patients and 3 of a total of 11 patient will reach day 100 after transplant without additional immunsuppressive drug treatment

SECONDARY OUTCOMES:
Overall Survival | day 100 after transplant
engraftment | day 100 after transplant
  absolute neutrophil count of > 0.5 x 10e9/l on 3 consecutive days
chimerism | day 100 after transplant
  Percentage of donor cells in leukocytes from peripheral blood or bone marrow
relapse incidence | day 100 after transplant
  cumulative incidence of relapse until day 100
acute GvHD | day 100 after transplant
  cumulative incidence of acute GvHD
non-relapse mortality | day 100 after transplant
  cumulative incidence of death from any cause without prior relapse or progression of malignant disease
immune reconstitution | day 100 after transplant
  relative and absolute counts of B- and T-lymphocyte subsets in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Scheid, MD PhD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany